CLINICAL TRIAL: NCT01976377
Title: Expression of Mucin Glycosylating Enzymes in Head and Neck Cancers and Its Correlation With Clinico-pathological Parameters.
Brief Title: Mucin Glycosylating Enzymes in Head and Neck Cancers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201307074RIND
Record Dates: First submitted 2013-10-22; First posted 2013-11-05 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Glycosyltion Enzymes and Function Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stage I, II, III, IV HNSCC: Stage I, II, III, IV HNSCC reveive treatment in NTUH

SUMMARY:
Head and neck squamous cell carcinoma(HNSCC) is the fourth common malignancy in Taiwan. It accounts for 5.8% of all cancers and causes 2,463 deaths per year. Aberrant glycosylation is the hallmark of most human cancers, including HNSCC, and affects many cellular properties. This study is aimed at exploring the role of mucin glycosylating enzymes in HNSCC.

DETAILED DESCRIPTION:
Glycosylation is the most common post-translational modification of proteins. Aberrant glycosylation is the hallmark of most human cancers and affect many cellular properties, including cell proliferation, apoptosis, differentiation, transformation, migration and immune response.

Though widely explored in various human cancers, the role of mucin glycosylating enzymes in HNSCC has not been elucidated. Our aims is to analyze the expression patterns of mucin glycosylating enzymes in HNSCC tissues. Furthermore, we will correlate the expression levels of mucin glycosylating enzymes with clinical characteristics of HNSCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer patients receiving operation in National Taiwan University Hospital

Exclusion Criteria:

* Recurrence or non-operable patients

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head and neck cancer patients receiving operation in National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Measure the expression of mucin glycosylating in head and neck cancer | 1~5 years after patient received surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jen Lou, M.D, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University, Taipei, Taiwan, Taiwan